CLINICAL TRIAL: NCT01318174
Title: Prevalence of Pulmonary Embolism in Exacerbations of Chronic Obstructive Pulmonary Disease
Brief Title: Pulmonary Embolism in Exacerbations of Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Sykehuset Innlandet HF (Other)
Responsible Party: Principal Investigator, Aleksander Talgøy Holten, MD, Sykehuset Innlandet HF
Other Study IDs: LE-KE
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Pulmonary Embolism; Chronic Obstructive Pulmonary Disease
Keywords: Pulmonary embolism; Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Embolism; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the prevalence of pulmonary embolism in our population of Chronic Obstructive Pulmonary Disease (COPD) patients admitted to hospital with dyspnea. The patients will undergo investigation for pulmonary embolism, according to current guidelines.

ELIGIBILITY:
Inclusion Criteria:

* known or suspected COPD
* COPD-exacerbation

Exclusion Criteria:

* other causes of dyspnea
* unable to perform CT pulmonary angio (contrast allergy, pregnancy)
* already included in the study (each patient included only once)
* use of anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known or suspected COPD admitted with an exacerbation of unknown aetiology
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of pulmonary embolism in exacerbations of COPD | one year

CONTACTS AND LOCATIONS:
Overall Officials: Aleksander T Holten, PhD, Principal Investigator — Sykehuset Innlandet HF
Locations (1):
- Sykehuset Innlandet, Lillehammer, Oppland, Norway